CLINICAL TRIAL: NCT07270965
Title: Understanding the Effect of Pre-Drying Moisturization on Skin Hydration
Brief Title: Moisturization and Skin Hydration Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Principal Investigator, Wingfield Rehmus, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H25-02646
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis (AD); Atopic Dermatitis (Eczema)
Keywords: Atopic Dermatitis; Eczema; AD; Moisturizer; Cream; Skin Hydration
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moisturizing while in shower/bath (Experimental)
  Interventions: Behavioral: Moisturizing while in shower/bath
- Moisturizing after towel drying (Experimental)
  Interventions: Behavioral: Moisturizing after towel drying

INTERVENTIONS:
Behavioral: Moisturizing while in shower/bath — Applying moisturizer in the shower/bath.
  Arms: Moisturizing while in shower/bath
Behavioral: Moisturizing after towel drying — Applying moisturizer out of the shower/bath after towel drying.
  Arms: Moisturizing after towel drying

SUMMARY:
Skin moisturization is important for patients with atopic dermatitis, commonly known as eczema. Moisturizing right after bathing is widely accepted as the best method to keep skin hydrated. However, there is conflicting research on the timing of moisturizing. The goal of this clinical study is to evaluate the preference of moisturizing while showering/bathing compared to after towel drying in adolescents aged 12-18 with eczema. The main question it aims to answer are:

* Which moisturization technique is preferred: while showering/bathing or after towel drying?
* How do these techniques affect investigator-assessed eczema severity, patient-reported itch scores, and objective skin hydration measurements?

Researchers will compare applying moisturizer while in the shower/bath to after towel drying and to which technique is preferred among participants and if there are different effects on eczema and skin hydration.

Participants will:

* Apply moisturizer while showering/bathing for one month and after towel drying for one month.
* Complete questionnaires on moisturization technique, skin feel, and itchiness.
* Undergo skin hydration measurements using a Corneometer® CM825 device.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of atopic dermatitis/eczema.
* Participants must be between the age of 12-18.
* Participants must be able to bathe independently.
* Participants will be English speaking and able to complete questionnaires.

Exclusion Criteria:

* Participants who use topical corticosteroids between one inch above the wrist and 1 inch below the elbow from 1 month on both arms prior to the study until the final visit.
* Participants who have a known allergy to the moisturizer cream (Cerave Moisturizing Cream) provided.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Preferring Each Moisturization Technique | Through study completion, an average of 2 months.
  Participant reported preference of moisturization technique

SECONDARY OUTCOMES:
Skin Hydration Level | Through study completion, an average of 2 months.
  Skin electrical capacitance measured using Corneometer® CM825 as an indicator of skin hydration.

OTHER OUTCOMES:
Eczema Severity Score | Through study completion, an average of 2 months.
  Eczema severity will be assessed by clinicians using the Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD™). Scores range from 1 to 4, with higher scores indicating more severe eczema/atopic dermatitis (worse outcome).
Itch Intensity | Through study completion, an average of 2 months.
  Itch intensity will be assessed using a patient-reported Numeric Rating Scale (NRS) ranging from 1 to 10, where higher scores indicate greater itch severity (worse outcome). Participants will report both average itch and worst itch experienced within the past 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, but aggregated data from all participants will be shared.